CLINICAL TRIAL: NCT03522155
Title: A Patient-Centered Approach to Integration of Life Expectancy Into Treatment Decision Making for Patients With Genitourinary Malignancy
Brief Title: Patient-Centered Communication of Life Expectancy Estimates in Genitourinary Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Timothy J. Daskivich, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00052777
Record Dates: First submitted 2018-04-18; First posted 2018-05-11 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer Stage I; Kidney Cancer Stage I; Bladder Cancer Stage II; Prostate Cancer Stage II
Keywords: Conjoint Analysis; Life Expectancy; Patient-centered
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial will involve two arms: (1) an intervention arm consisting of a patient-centered communication strategy for life expectancy and (2) standard of care treatment counseling. The intervention will be randomized at the level of the patient to balance study arms in terms of measured and unmeasured patient characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Intervention: (1) Subjects will be provided with patient-specific LE estimates, (2) counseling physicians will receive "talking points" to assist in meaningful communication of life expectancy, and (3) subjects will complete a computer-based conjoint analysis exercise prior to counseling.
  Interventions: Behavioral: Patient-centered communication of life expectancy
- Standard-of-care Arm (No Intervention): Patients in the standard-of-care arm will not receive an intervention and will receive the usual standard of care for treatment counseling.

INTERVENTIONS:
Behavioral: Patient-centered communication of life expectancy — The intervention arm will test if patient-specific LE estimates via a targeted, patient-centered communication approach paired with LE-specific conjoint analysis data improves decisional conflict, quality of LE discussion, and reduces rates of overtreatment of Genitourinary malignancies.
  Arms: Intervention Arm

SUMMARY:
Investigators will conduct a randomized trial to determine if providing patient-specific life expectancy estimates during treatment counseling via a targeted, patient-centered communication approach improves shared decision making and reduces rates of overtreatment of genitourinary malignancies.

DETAILED DESCRIPTION:
Subjects in the intervention arm will be provided with life expectancy estimates specific to their age and health status. Life expectancy estimates for prostate and kidney cancer patients will be estimated by age and Charlson comorbidity score cutoffs, and life expectancy for bladder cancer patients will be determined using definitions as noted by Cho et al. Talking points will be provided to counseling physicians on how to meaningfully communicate life expectancy data. Subjects will also complete a computer-based conjoint analysis exercise prior to the counseling visit; results will be used to help physicians understand how the subject values life expectancy compared with other decision attributes. The control arm will consist of the current standard of care for treatment counseling.

The intervention will be randomized at the level of the patient after stratification by type of cancer.

All participants will be asked to fill out a validated questionnaire to measure decisional conflict at the conclusion of their counseling visit. Investigators will audiotape treatment counseling visits to allow for qualitative analysis of the quality of communication of life expectancy information. Treatment choice will be documented to assess rates of aggressive versus non-aggressive treatment among patients with limited life expectancy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed clinical T1-2 prostate adenocarcinoma with Gleason scores of 7 or less
* Newly diagnosed clinical T1a kidney cancer or renal masses < 4cm
* Newly diagnosed clinical T2 nonmetastatic urothelial carcinoma of the bladder

Exclusion Criteria:

* Under 18 years of age
* Subjects with difficulty communicating or dementia
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict | At time of treatment decision, up to 12 weeks after diagnosis
  Decisional conflict evaluated based on the total decisional conflict score (DCS). The scale measures the degree of certainty/uncertainty an individual feels in selecting choices, feelings of being uninformed or unclear about values, and feelings of satisfaction with the selected decision. Scores range from 0 to 100. A total score of 0 indicates no decisional conflict, while a score of 100 indicates extremely high levels of decisional conflict.

SECONDARY OUTCOMES:
Treatment Choice | At time of treatment decision, up to 12 weeks after diagnosis
  The investigator will look at the difference in odds of aggressive vs. non-aggressive treatment. Aggressive treatment will be defined as surgery, radiation or ablative therapy; non-aggressive treatment will be defined as active surveillance, watchful waiting, or medical management.
Mention of life expectancy | At time of treatment decision, up to 12 weeks after diagnosis
  Difference in odds of mention of life expectancy (binary variable)
Time devoted to life expectancy | At time of treatment decision, up to 12 weeks after diagnosis
  Difference in proportion of time devoted to discussion of life expectancy (minutes discussed/total minutes)
Number of questions asked about life expectancy | At time of treatment decision, up to 12 weeks after diagnosis
  Difference in number of questions asked about life expectancy

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Daskivich, MD, MSHPM, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Investigators on this project will follow the NIH Grants Policy Statement concerning the sharing of research data and will make available to the public the results of the collaborative research and any accompanying data supported by this grant if funded. Such data shall be available in a timely fashion to researchers and/or the public upon request, provided that (1) such data may not be available until the time that it is used in connection with publication(s), (2) such data may be withheld for a reasonable amount of time to evaluate the impact of disclosure on patentability consistent with the Bayh-Dole Act, and (3) such data will not include any information that could be used to identify individual participants.

REFERENCES:
- [Background] Daskivich TJ, Tan HJ, Litwin MS, Hu JC. Life Expectancy and Variation in Treatment for Early Stage Kidney Cancer. J Urol. 2016 Sep;196(3):672-7. doi: 10.1016/j.juro.2016.03.133. Epub 2016 Mar 21. PMID 27012644
- [Background] Daskivich TJ, Lai J, Dick AW, Setodji CM, Hanley JM, Litwin MS, Saigal C; Urologic Diseases in America Project. Variation in treatment associated with life expectancy in a population-based cohort of men with early-stage prostate cancer. Cancer. 2014 Dec 1;120(23):3642-50. doi: 10.1002/cncr.28926. Epub 2014 Jul 17. PMID 25042117
- [Background] Cho H, Klabunde CN, Yabroff KR, Wang Z, Meekins A, Lansdorp-Vogelaar I, Mariotto AB. Comorbidity-adjusted life expectancy: a new tool to inform recommendations for optimal screening strategies. Ann Intern Med. 2013 Nov 19;159(10):667-76. doi: 10.7326/0003-4819-159-10-201311190-00005. PMID 24247672
- [Background] Ryan M, Farrar S. Using conjoint analysis to elicit preferences for health care. BMJ. 2000 Jun 3;320(7248):1530-3. doi: 10.1136/bmj.320.7248.1530. No abstract available. PMID 10834905
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294